CLINICAL TRIAL: NCT06989593
Title: Breaking Silence Through Story: A Narrative Medicine Intervention for Parents of Children With Urogenital Conditions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sarah Schlegel (Other)
Collaborators: Harvard Catalyst Pilot Grant (Unknown)
Responsible Party: Sponsor-Investigator, Sarah Schlegel, Attending Physician in Endocrinology, Instructor of Pediatrics, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-P00051291; 89676 (Other Grant/Funding Number: Harvard Catalyst Pediatric Clinical Research Pilot Grant)
Record Dates: First submitted 2025-05-22; First posted 2025-05-25 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-05

CONDITIONS: DSD; Hypospadias
Keywords: Disorders of Sex Development; Hypospadias; Anxiety; Stress, Psychological; Parents; Psychological Adaptation; Writing; Narrative Therapy; Qualitative Research; Patient Participation; Social Support; Mental Health; Interpersonal Relations; Parent-Child Relations; Urogenital Abnormalities; Female Urogenital Diseases; Urogenital Diseases; Penile Diseases; Genital Diseases, Male; Genital Diseases; Male Urogenital Diseases; Congenital Abnormalities; Gonadal Disorders; Endocrine System Diseases
MeSH Terms: conditions — Hypospadias; Disorders of Sex Development; Anxiety Disorders; Stress, Psychological; Patient Participation; Psychological Well-Being; Urogenital Abnormalities; Female Urogenital Diseases; Urogenital Diseases; Penile Diseases; Genital Diseases, Male; Genital Diseases; Male Urogenital Diseases; Congenital Abnormalities; Gonadal Disorders; Endocrine System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Narrative Medicine Journaling Intervention (Experimental): All participants in this single-arm pilot study will complete baseline GAD-7 anxiety assessments, participate in a guided journaling program, complete follow-up GAD-7 assessments, and take part in a qualitative interview. Parents of children with urogenital conditions (differences of sex development and hypospadias) will receive the narrative medicine intervention over a period of several weeks, with pre- and post-intervention anxiety measurements and interview assessments.
  Interventions: Behavioral: Narrative Medicine Journaling Intervention

INTERVENTIONS:
Behavioral: Narrative Medicine Journaling Intervention — Participants will complete the GAD-7 anxiety assessment at baseline. They will then receive a physical journal containing 5 structured, therapeutic writing prompts designed to help process emotions related to their child's diagnosis. Prompts focus on processing experiences with diagnosis, addressing uncertainty, coping with stigma, and developing resilience. Parents will be instructed to complete the 5 journal entries, spending 15-20 minutes on each writing session at least once per week. Following completion of the journaling intervention, participants will complete a follow-up GAD-7 assessment and take part in a 30-45 minute qualitative interview to further assess perceived changes in anxiety, stress, and coping strategies, and to gather feedback on potential group-based writing programs.
  Other Names: Therapeutic Writing; Reflective Journaling; Guided Narrative Intervention; Narrative Medicine

SUMMARY:
The goal of this clinical trial is to learn whether a journaling intervention can reduce stress and anxiety in parents of children with urogenital conditions (such as differences of sex development and hypospadias).

The main questions it aims to answer are:

* Does guided journaling help to reduce anxiety levels in parents of children with urogenital conditions?
* What are parents' perspectives on group-based writing interventions for future support programs?

Participants will:

* Complete a short anxiety questionnaire (the General Anxiety Disorder-7 scale) at the beginning of the study
* Receive a physical journal with 5 writing prompts designed to help process emotions related to their child's condition
* Complete 5 journal entries over several weeks, writing about their experiences and feelings
* Complete the same anxiety questionnaire again after finishing the journal entries
* Participate in a 45-minute interview to discuss how the journaling affected their stress levels and gather feedback on potential group-based writing programs

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian of a child (age 0-17 years) diagnosed with a urogenital condition (differences of sex development and/or hypospadias)
* Able to read and understand English
* Child receives care at Boston Children's Hospital
* Willing to complete a guided journaling intervention (through writing or dictation) over a period of approximately 5 weeks
* Willing to participate in a 45 minute follow-up interview
* Able to provide informed consent

Exclusion Criteria:

* Parent/guardian with severe psychiatric disorder that would interfere with participation as determined by referring physician
* Parent/guardian unable to complete either written journaling activities or dictation
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in GAD-7 Anxiety Scores | Change from baseline (pre-intervention) to approximately 6 weeks post-intervention initiation
  Change from baseline in General Anxiety Disorder-7 (GAD-7) scores. The GAD-7 is a validated 7-item self-report questionnaire used to assess anxiety symptom severity. Scores range from 0-21, with higher scores indicating greater anxiety symptoms.

SECONDARY OUTCOMES:
Qualitative Assessment of Anxiety Related to Child's Diagnosis | Measured at one follow-up interview, approximately 6 weeks after intervention initiation
  Semi-structured interviews to assess participants' self-reported changes in anxiety specifically related to their child's urogenital condition following the narrative medicine intervention, including perceived changes in stress, worry frequency, and emotional distress related to the diagnosis.
Changes in Parental Coping Strategies | Measured at one follow-up interview, approximately 6 weeks after intervention initiation
  Qualitative assessment through semi-structured interviews of participants' self-reported changes in coping mechanisms, including reduction in feelings of self-blame, increased sense of control, and development of new strategies for managing uncertainty following the journaling intervention.
Interest in Group-Based Writing Interventions | Approximately 6 weeks after intervention initiation
  Assessment of parents' interest in and preferences for potential group-based writing interventions, including identification of perceived benefits, potential barriers to participation, and suggestions for implementation approaches. Measured at one follow-up interview, approximately 6 weeks after intervention initiation
Feasibility and Acceptability of Journaling Intervention | Approximately 6 weeks after intervention initiation
  Assessment of participation rates, completion of journal entries, and participant feedback on the structure, content, and delivery of the journaling intervention to inform future program development. Measured at one follow-up interview, approximately 6 weeks after intervention initiation

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this pilot study primarily collects sensitive qualitative data through personal narratives and interviews concerning parents' experiences with their children's urogenital conditions. The small sample size and detailed personal accounts could potentially lead to participant identification even if de-identified, raising significant confidentiality and privacy concerns. Additionally, during the informed consent process, participants will not have been specifically asked for permission to share their raw data beyond the research team. The study will instead focus on sharing aggregate findings and thematic analyses while protecting participants' confidentiality. If future researchers are interested in the data, specific requests may be considered by the IRB on a case-by-case basis with appropriate data use agreements.